CLINICAL TRIAL: NCT06723860
Title: The Critical Care Recovery Program: Use of a Structured Clinic Visit to Reduce Adverse Drug Events in ICU Survivors
Acronym: CCRP
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Marnie Wilson, Clinical Assistant Professor of Medicine, University of British Columbia
Other Study IDs: H24-03124
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Post Intensive Care Syndrome (PICS); Polypharmacy; Adverse Drug Events; Critical Care, Intensive Care
MeSH Terms: conditions — postintensive care syndrome; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective control cohort: Retrospectively collected data on a group of intensive care survivors who were not referred for a post-ICU clinic visit.
- Intervention cohort: Patients meeting FICM criteria who are referred for a CCRP clinic visit and consent to participation in research

SUMMARY:
Background and Objective: Intensive Care Units (ICUs) save lives, but many ICU survivors face ongoing health issues, including adverse drug events (ADEs) from medications started during their hospital stay. These ADEs lead to emergency department visits and hospital admissions. Our project aims to improve the health of ICU survivors by creating a clinic that focuses on managing post-ICU health. The clinic will track and address medical issues that arise after ICU discharge and focus on deprescribing, or safely stopping, medications that may no longer be needed or could be harmful.

Project Plan: The clinic will be set up within the CARES clinic at VGH. Patients will be enrolled when they leave the ICU and will have follow up visits after hospital discharge. During these visits, the team will review each patient's medications and develop a personalized plan to reduce or stop unnecessary medications. We will also monitor patients for any new health issues that arise and provide eduction to patients and caregivers about managing their health.

Research and Evaluation: We will collect and analyze data on patient health outcomes, including the incidence of ADEs, hospital reeadmissions, and emergency department visits. We hope to show that patients who receive follow up care have better health outcomes and use fewer healthcare resources than a historical cohort. This data will help us demonstrate the cost-effectiveness of the clinic and support the need for expanding ICU follow up programs in British Columbia.

Long-term goals: We plan to establish a post-ICU care working group and expand the clinic model to other hospitals. Over the long term, we hope to standardize post-ICU care across BC, ensuring that all ICU survivors have access to comprehensive follow up care. This project will also lay the groundwork for future research on deprescribing medications for ICU related complications, which tend to improve or resolve once critical illness has resolved. The CCRP clinic will provide a setting to conduct clinical deprescription trials to establish whether long-term treatment of these complications is necessary.

Conclusion: Establishing a post-ICU discharge follow up clinic with a focus on deprescription has the potential to improve the long-term health and quality of life for ICU survivors. By reducing unnecessary medications, we can prevent complications, reduce hospital readmissions and demonstrate the value of comprehensive post-ICU follow up care.

ELIGIBILITY:
Inclusion Criteria:

* Patient being discharged to ward, home or repatriated to local health centre AND ONE OR MORE OF

  * Duration of mechanical ventilation >72 hours
  * Length of stay in critical care >96 hours
  * Out of hospital arrest
  * Maternal critical illness
  * Trauma
  * Significant ICU delirium
  * Unexpected adverse outcomes of planned treatment

Exclusion Criteria:

* Patient discharged for palliative care or expected to die within the next two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting inclusion / exclusion criteria above (per FICM guidelines for critical care recovery program follow up)
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital in the year following hospital discharge | 1 year

SECONDARY OUTCOMES:
Emergency department visits and hospital admissions in the year following ICU admission | 1 year

IPD SHARING:
Plan to Share IPD: Yes
Data will be retained in a database for as long as the clinic is active. Other researchers with REB approval may request access to the data, which will be long term ICU follow up data and potentially applicable to many other studies. This data can be released at the discretion of the principal investigator.